CLINICAL TRIAL: NCT03890874
Title: An Analysis of the Efficacy of Different Teaching Modalities in Imparting Adult CPR Skills in First Year Medical Students
Brief Title: An Analysis of the Efficacy of Different Teaching Modalities
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Appu Suseel, Assistant Professor, Jubilee Mission Medical College and Research Institute
Other Study IDs: 18/19/IEC/JMMC&RI; U1111-1229-7995 (Other: World Health Organisation)
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Simulation Training
Keywords: Cardiopulmonary Resuscitation; Teaching techniques; Basic Life Support training; Simulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First year medical students: First year medical students of jubilee mission medical college and research institute

SUMMARY:
Didactic lectures are the currently used mode of imparting training to medical students. Use of other modes of teaching like simulation is still in its infancy. Simulation, as a teaching tool may aid in longer retention of the learning contents and also provides a safe environment for the students to practice their skills after knowledge acquisition. The aim of the study is to analyze the efficacy of different teaching modalities in imparting a particular skill, namely adult cardiopulmonary resuscitation (CPR) which is a life saving skill in first year medical students. The study population includes all the first year MBBS students and the duration of the study is 1 month. A clarity as to which mode of teaching will be ideal for memory retention is the expected outcome of this study.

DETAILED DESCRIPTION:
Introduction

Our current medical curriculum devotes a large percentage of its time to knowledge acquisition by means of didactic lectures. Psychomotor skill acquisition takes a back seat. Certain lifesaving skills like basic life support skill training have not even made an appearance in the current curriculum. Equal time distribution to cognitive and psychomotor skills should be allotted for a subject as practical as MBBS .Simulation can prove to be a valuable tool in imparting skill training. The present study aims to evaluate the efficacy of different teaching modalities in imparting lifesaving skills in first year MBBS students.

Methods

This Cross sectional study is conducted among 33 first year students who consented to participate. Institutional ethics clearance was also obtained. The students were divided into three groups, each undergoing didactic lecture, animation based videos and simulation studies. Pretest, posttest and skills test was administered to them. One way anova, Paired t test were some of the statistical test employed using SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* All First year MBBS Students who are willing to participate

Exclusion Criteria:

* Prior training in adult CPR skills
* Physical disabilities that does not permit performing high quality CPR

Ages: 18 Years to 20 Years | Sex: All
Age Groups: Adult
Study Population: First year Medical students of Jubilee Mission Medical college and Research Institute.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-17 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
comparing the mean post test score of groups of students that underwent training using different teaching modalities assessed using a ten part multiple choice questionnaire. | 4 hours
  Amongst visual, didactic and simulation models of teaching, to identify the more effective strategy to impart Basic Life Support (BLS) knowledge to first year medical students through a four hour training programme, by comparing the mean post test scores of each group

SECONDARY OUTCOMES:
comparing the change in the baseline test score amongst first year medical students taught by visual, didactic and simulation models. | 4 hours
  students through a four hour training programme, by comparing the mean pre test and post test scores of each group
comparing the mean score of groups of students that underwent training using different teaching modalities, assessed by an examiner testing their skills using a pre set basic life support checklist proforma. | 4 hours
  comparing the effectiveness of each teaching modality amongst first year medical students to impart Adult Cardiopulmonary Resuscitation (CPR) skills assessed by an examiner observing and testing their skills using a pre set checklist proforma.

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi Panchu, MD, Study Chair — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee mission medical college and research institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: No